CLINICAL TRIAL: NCT04944472
Title: Opportunities for the Perception of Information on the Primary Prevention of Cardiovascular Diseases in Persons Suffering From Hypertension Through the Social Network Instagram
Brief Title: Possibilities of Perceiving Information on the Primary Prevention of Cardiovascular Diseases in Persons Suffering From Essential Hypertension Through a Social Network
Acronym: SocialCor
Status: Completed | Type: Observational
Sponsor: Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/1
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Prevention, Arterial Hypertension
Keywords: digital prevention, primary prevention, secondary prevention, hypertension, patient education, social media
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group I: All participants will be divided into 4 groups (4 separate accounts), similar in gender, age and social status:
  in group I, project participants will only be presented with video publications on each of the declared topics (8 in total).
  Interventions: Behavioral: HDKQ questionnaire
- group II: All participants will be divided into 4 groups (4 separate accounts), similar in gender, age and social status:
  in group II - only text publications (total 8).
  Interventions: Behavioral: HDKQ questionnaire
- group III: All participants will be divided into 4 groups (4 separate accounts), similar in gender, age and social status:
  in group III - first text publications, and then video publications (16 in total).
  Interventions: Behavioral: HDKQ questionnaire
- group IV: All participants will be divided into 4 groups (4 separate accounts), similar in gender, age and social status:
  in group IV - first video publications, and then text publications (16 in total).

INTERVENTIONS:
Behavioral: HDKQ questionnaire — Studying the possibilities of perceiving information on the primary prevention of cardiovascular diseases in persons suffering from hypertension through the social network Instagram
  Groups: group I; group II; group III

SUMMARY:
A randomized, prospective study conducted on the basis of a social network (Instagram platform), two-stage. At the first stage, the online school "Save Your Heart" was announced and 945 applicants were enrolled in the training. The online school curriculum consisted of the following blocks: "Risk Factors for Cardiovascular Diseases (CVD)", "Healthy Nutrition for the Heart", "Cholesterol. What is important for the patient to know? "," Physical activity for the prevention of CVD "," Overweight and obesity "," Smoking as a risk factor for CVD "," AH: diagnosis "," AH: treatment "," Myocardial infarction: diagnosis and treatment". At the 2nd stage, 125 participants were selected by random randomization, then distributed into 4 training groups to provide training materials: group 1 (n = 31) - then text publications up to 4 thousand characters, group 2 (n = 31) - short video clips up to 5 minutes, group 3 (n = 33) - first text publications, then video clips, group 4 (n = 30) - video clips, then text publications. Before and after school, respondents from all four groups completed the HDKQ questionnaire.

DETAILED DESCRIPTION:
To study the potential of the Instagram social network in increasing the medical literacy of people with essential hypertension and to develop methodological approaches to informing the population about the primary prevention of cardiovascular diseases through social networks, including hypertension.

1. To assess the level of knowledge about risk factors and cardiovascular diseases among users of social networks with essential hypertension.
2. Conduct a comparative assessment of the impact of the type of information materials for patients in social networks (Group I - text, Group II - video, Group III - video + text, Group IV - text + video) on the level of its understanding and assimilation by persons with essential hypertension.
3. To study the possibilities of perceiving information on the primary prevention of cardiovascular diseases, depending on the gender, age and social status of users of social networks suffering from hypertension.

The research site is the social network Instagram, 4 new accounts will be created to complete the assigned tasks.

An adapted HDKQ (Heart Disease Knowledge Questionnaire) with additional gender, age and social status questions will be sent to those eligible for inclusion before the start of the educational program. Respondents to the questions of the questionnaire should be sent in text format to the private messages of the project account.

The format of interaction with the audience includes 8 text publications up to 4 thousand characters and 8 video publications up to 5 minutes long.

Text and video publications will be identical in terms of text content, and they will also reflect the answers to each question of the HDKQ questionnaire.

Publication topics:

1. Risk factors for cardiovascular disease.
2. Healthy food for the heart.
3. "Good" and "bad" cholesterol. What is important to know?
4. Physical activity. How much movement does it take to keep your heart healthy?
5. Overweight and obesity.
6. Smoking as a risk factor for cardiovascular diseases.
7. Hypertension: diagnosis, treatment goals.
8. Myocardial infarction is one of the most formidable cardiovascular complications.

All participants will be divided into 4 groups (4 separate accounts), similar in gender, age and social status:

in group I, project participants will only be presented with video publications on each of the declared topics (8 in total), in group II - only text publications (total 8), in group III - first text publications, and then video publications (16 in total), in group IV - first video publications, and then text publications (16 in total).

Upon completion of the educational program, participants will again be asked to answer the questions of the adapted HDKQ (Heart Disease Knowledge Questionnaire) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of arterial hypertension
2. Informed consent signed by the respondent.

Exclusion Criteria:

1. No diagnosis of arterial hypertension

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The total number of people who listened to and read the material of the online school was 2108 people, the total involvement (comments, reposts, saving the material) was 1598 people. The average percentage of watching videos is 22%. The audience of the online school is mostly female (84%), with an average age of 45.9 ± 12.3 years. 80.8% of the participants had higher than secondary education.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Awareness of risk factors for arterial hypertension as measured by the HDKQ questionnaire | Before and after school

CONTACTS AND LOCATIONS:
Overall Officials: S. P. Morozov, Study Director — Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department; A. V. Vladzymyrskyy, Study Director — Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Locations (1):
- Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No